CLINICAL TRIAL: NCT00640796
Title: Pilot Study of Expanded, Activated Haploidentical Natural Killer Cell Infusions for Non-B Lineage Hematologic Malignancies and Solid Tumors
Brief Title: Pilot Study of Expanded, Donor Natural Killer Cell Infusions for Refractory Non-B Lineage Hematologic Malignancies and Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Assisi Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKEXP; R01CA113482 (NIH)
Record Dates: First submitted 2008-03-14; First posted 2008-03-21 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Acute, T-Cell; Juvenile Myelomonocytic Leukemia Lymphoblastic; T-cell Lymphoblastic Lymphoma; Myelodysplastic Syndrome
Keywords: Hematologic malignancies, non-B lineage; NK cell expansion; CliniMACS device; Immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Hematologic Neoplasms | interventions — Drug Therapy; Cyclophosphamide; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Participants undergo haploidentical donor derived natural killer cell infusion (cells obtained from donors and selected using CliniMACS cell selection system) and chemotherapy (cyclophosphamide, fludarabine, interleukin-2, mesna).
  Interventions: Procedure: Haploidentical donor derived natural killer cell infusion; Drug: Chemotherapy; Device: CliniMACS

INTERVENTIONS:
Procedure: Haploidentical donor derived natural killer cell infusion — Therapeutic cell infusion
Drug: Chemotherapy — Cyclophosphamide, Fludarabine, Interleukin-2, Mesna
  Other Names: cyclophosphamide: cytoxan; fludarabine: Fludara(R); interleukin-2: IL-2, aldesleukin, Proleukin(R); mesna: Mesnex(R)
Device: CliniMACS — Cell selection system based on magnetic-activated cell sorting

SUMMARY:
Modern frontline therapy for patients with hematologic malignancies is based on intensive administration of multiple drugs. In patients with relapsed disease, response to the same drugs is generally poor, and dosages cannot be further increased without unacceptable toxicities. For most patients, particularly those who relapse while still receiving frontline therapy, the only therapeutic option is hematopoietic stem cell transplantation (SCT). For those who relapse after transplant, or who are not eligible for transplant because of persistent disease, there is no proven curative therapy.

There is mounting evidence that NK cells have powerful anti-leukemia activity. In patients undergoing allogeneic SCT, several studies have demonstrated NK-mediated anti-leukemic activity. NK cell infusions in patients with primary refractory or multiple-relapsed leukemia have been shown to be well tolerated and void of graft-versus-host disease (GVHD) effects. Myeloid leukemias are particularly sensitive to NK cells cytotoxicity, while B-lineage acute lymphoblastic leukemia (ALL) cells are often NK-resistant. We have developed a novel method to expand NK cells and enhance their cytotoxicity. Expanded and activated donor NK cells have shown powerful anti-leukemic activity against acute myeloid leukemia (AML) cells and T-lineage ALL cells in vitro and in animal models of leukemia.

The present study represents the translation of these laboratory findings into clinical application.We propose to determine the safety of infusing expanded NK cells in pediatric patients who have chemotherapy refractory or relapse hematologic malignancies including AML, T-lineage ALL, T-cell lymphoblastic lymphoma (T-LL), chronic myelogenous leukemia (CML), juvenile myelomonocytic leukemia (JMML),myelodysplastic syndrome (MDS), Ewing sarcoma family of tumors (ESFT) and rhabdomyosarcoma (RMS). The NK cells used for this study will be obtained from the patient's family member who will be a partial match to the patient's immune type (HLA type).

DETAILED DESCRIPTION:
Secondary objectives include the evaluation of the in vivo lifespan and phenotype of the expanded NK cells and explore the efficacy of these donor NK cells in study participants with relapsed or refractory hematologic malignancies or sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 18 years of age (may be greater than 18 years of age if currently a St. Jude patient).
* Patients with relapsed or refractory AML, T-ALL/T-LL, mixed lineage leukemia, CML, JMML, MDS, ESFT or RMS who are not eligible for SCT and have persistent disease after remission induction(s) therapy as evidenced by bone marrow morphology, cytogenetics, flow cytometry, molecular pathology, and/or restaging scans.
* At least two weeks since receipt of any biological therapy, systemic chemotherapy, and/or radiation therapy.
* Shortening fraction greater than or equal to 25%.
* Creatinine clearance or glomerular filtration rate greater than or equal to 50 cc/min/1.73 m^2.
* Pulse oximetry greater than or equal to 92% on room air.
* Direct bilirubin less than or equal to 3.0 mg/dL.
* Karnofsky or Lansky performance score of greater than or equal to 50.
* No known allergy to murine products or HAMA testing results within normal limits.
* Does not have a current pleural or pericardial effusion.
* Has a suitable adult family member donor available for NK cell donation.
* Is not receiving more than the equivalent of prednisone 10 mg daily.
* Not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).
* Not breast feeding.

Eligibility criteria prior to initiation of protocol therapy (preparative regimen)

* Alanine aminotransferase (ALT) is no more than 2 times the upper limit of normal.
* Aspartate transaminase (AST) is no more than 2 times the upper limit of normal.
* Has recovered from all acute NCI Common Toxicity Criteria grade II-IV non-hematologic acute toxicities resulting from prior therapy per the judgment of the principal investigator

Eligibility criteria (NK cell DONOR):

* Family member with a greater than or equal to 3 of 6 HLA match to recipient.
* At least 18 years of age.
* HIV negative.
* Not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).
* Not breast feeding.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2008-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of expanded NK cells in research participants with relapsed or refractory hematologic malignancies and sarcomas. | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: David Shook, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org